CLINICAL TRIAL: NCT03161080
Title: Effect of Single Instillation of Three Different Topical Lubricants on Tear Film Thickness in Patients With Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-250716
Record Dates: First submitted 2017-03-28; First posted 2017-05-19 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry Eye Neovis (Experimental): 20 Patients with dry eye syndrome receiving Neovis Total Multi Eyedrops
  Interventions: Device: Neovis Total Multi® Eye Drops
- Dry Eye Vismed (Experimental): 20 Patients with dry eye syndrome receiving Vismed Multi Eyedrops
  Interventions: Device: Vismed Multi® Eye Drops
- Dry Eye Hydrabak (Experimental): 20 Patients with dry eye syndrome receiving Hydrabak Eyedrops
  Interventions: Device: Hydrabak® Eye Drops

INTERVENTIONS:
Device: Neovis Total Multi® Eye Drops — Eye Drops containing Sodium hyaluronate (0.18%), lipoic acid, hydroxypropyl methylcellulose
  Arms: Dry Eye Neovis
Device: Vismed Multi® Eye Drops — Eye Drops containing Sodium hyaluronate (0.18%), potassium chloride, disodium phosphate
  Arms: Dry Eye Vismed
Device: Hydrabak® Eye Drops — Eye Drops containing sodium chloride (0,9%), sodium dihydrogen phosphate dehydrate
  Arms: Dry Eye Hydrabak

SUMMARY:
The prevalence and incidence of dry eye syndrome (DES) is constantly increasing. Several therapeutic strategies have been proposed, but still no ideal regimen has been found. Recently, a new method for the non- invasive measurement of tear film thickness (TFT) based on optical coherence tomography (OCT) has been developed. It has been shown in previous studies that TFT correlates well with objective signs as well as with subjective symptoms of DES.

In the present study the effects of three different topical lubricants (Neovis total multi®, Vismed multi® and Hydrabak® eye drops) on tear film thickness in patients with moderate to severe DES will be investigated using this device.

Tear film thickness will be measured at baseline and at defined time points after single instillation. The course of tear film thickness during this study day will provide information about the corneal residency time of the three different eye drops. Patients with moderate to severe DES will be randomized to receive either Neovis total multi®, Vismed multi® or Hydrabak® eye drops. Assessment of lipid layer thickness of the tear film will be performed before and at pre-specified time points after instillation as secondary outcome.

Other clinical measures for DES such as determination of tear film break up time (TFBUT), corneal fluorescein staining, Schirmer I test and subjective assessments will also be performed.

ELIGIBILITY:
Inclusion Criteria

Patients will be eligible for inclusion if all these criteria are respected:

1. Age of at least 18 years
2. Provides written informed consent prior to study-related procedures at the screening visit
3. Is able to understand and willing to comply with the procedures and the actions asked of him/her
4. History of dry eye syndrome for at least 3 months
5. Reports at least 2 of the following symptoms related to dry eye syndrome: foreign body sensation, pain, itching, stinging, epiphora, photophobia or blurred vision
6. Tear Break Up Time (BUT) ≤ 10 seconds or Schirmer I test ≤ 10 mm
7. OSDI score ≥ 23 points
8. Normal ophthalmic findings except dry eye syndrome

Exclusion Criteria

Patients will be excluded under the following circumstances:

1. Participation in a clinical trial in the 3 weeks preceding the study
2. Symptoms of a clinically relevant illness in the 3 weeks before the first study day
3. Presence or history of a severe medical condition as judged by the clinical investigator
4. Intake of parasympathomimetic or anti-psychotic drugs
5. Wearing of contact lenses
6. Glaucoma in the medical history
7. Treatment with corticosteroids in the 4 weeks preceding the study
8. Topical treatment with any ophthalmic drug except topical lubricants in the 4 weeks preceding the study
9. Ocular infection or clinically significant inflammation not related to dry eye syndrome
10. Ocular surgery in the 3 months preceding the study
11. Sjögren's syndrome
12. Stevens-Johnson syndrome
13. History of allergic conjunctivitis
14. Pregnancy, planned pregnancy or lactating
15. Known hypersensitivity to any component of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Change in tear film thickness | 1 day
  Change in tear film thickness measured with optical coherence tomography (OCT) at predose and at defined time points after instillation of eyedrops

SECONDARY OUTCOMES:
Change in lipid layer thickness | 1 day
  Change in lipid layer thickness measured with the LipiViewII Ocular Surface Interferometer at predose and at defined time points after instillation of eyedrops
Tear Break Up Time (TBUT) | 2 weeks
  Tear Break Up Time measured at screening visit and on study day
Visual Analogue Scale (VAS) | 2 weeks
  Visual Analogue Scale about dry eye symptoms at screening visit and on study day
Schirmer I test | 2 weeks
  Schirmer I test measured at screening visit and on study
Ocular Surface Disease Index (OSDI) score | 1 day
  Ocular Surface Disease Index (OSDI) score assessed with questionnaire at screening visit
Corneal fluorescein staining | 2 weeks
  Corneal fluorescein staining at screening visit and on study day
Visual acuity | 2 weeks
  Visual acuity assessed at screening visit and on study day
Intraocular pressure (IOP) | 1 day
  Intraocular pressure measured at screening visit

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Szegedi S, Scheschy U, Schmidl D, Aranha Dos Santos V, Stegmann H, Adzhemian N, Fondi K, Bata AM, Werkmeister RM, Couderc C, Schmetterer L, Garhofer G. Effect of Single Instillation of Two Hyaluronic Acid-Based Topical Lubricants on Tear Film Thickness in Patients with Dry Eye Syndrome. J Ocul Pharmacol Ther. 2018 Nov;34(9):605-611. doi: 10.1089/jop.2018.0069. Epub 2018 Oct 16. PMID 30325687